CLINICAL TRIAL: NCT00371215
Title: A Phase 2 Study of Recombinant Human Thrombin (rThrombin) Administered Using a Spray Applicator in Subjects Undergoing Autologous Skin Grafting Following Burn or Traumatic Skin Injury
Brief Title: Study of Recombinant Human Thrombin for Bleeding During Autologous Skin Grafting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Allan Alexander, MD, ZymoGenetics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 499E02
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Surgical Hemostasis
Keywords: hemostasis; grafting, skin; hemostatics; phase 2
MeSH Terms: interventions — recombinant human thrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): rThrombin
  Interventions: Biological: rThrombin

INTERVENTIONS:
Biological: rThrombin — 1000 U/mL applied topically

SUMMARY:
The purpose of this study is to evaluate whether rThrombin is safe when used for controlling bleeding during skin graft surgery.

DETAILED DESCRIPTION:
This is a Phase 2 multiple site, single-arm, open-label study designed to evaluate the safety of rThrombin in subjects of age 2 to 75 years who are receiving a partial- or full-thickness autologous sheet or mesh grafts following burn or traumatic skin injury. After establishing eligibility, study participants will be treated with topical spray rThrombin at the skin graft recipient site during autologous skin graft surgery. There will be a 1-month follow-up period after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Autologous skin grafting with sheet or mesh grafts following burn or traumatic skin injury

Exclusion Criteria:

* Known antibodies or hypersensitivity to thrombin or other coagulation factors

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | Up to day 29

SECONDARY OUTCOMES:
The incidence and grade of clinical laboratory abnormalities | Up to day 29
The incidence of anti-rThrombin product antibodies | Up to day 29
The incidence of hemostasis | Up to 20 minutes
The percentage of graft take | Up to day 29
The incidence of re-grafting | Up to day 29

CONTACTS AND LOCATIONS:
Overall Officials: Allan Alexander, MD, Study Director — ZymoGenetics
Locations (1):
- Richard M. Fairbanks Burn Center, Wishard Hospital, Indianapolis, Indiana, United States